CLINICAL TRIAL: NCT01373073
Title: Evaluation of a Novel Human Milk Fortifier in Preterm Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK37
Record Dates: First submitted 2011-06-08; First posted 2011-06-14 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Preterm Infants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Human Milk Fortifier (Experimental): Experimental human milk fortifier to be added to human milk
  Interventions: Other: Experimental human milk fortifier
- Control Human Milk Fortifier (Active Comparator): Control human milk fortifier to be added to human milk
  Interventions: Other: Control human milk fortifier

INTERVENTIONS:
Other: Experimental human milk fortifier — Human milk fortifier to be added to human milk feedings
  Arms: Experimental Human Milk Fortifier
Other: Control human milk fortifier — Control human milk fortifier to be added to human milk
  Arms: Control Human Milk Fortifier

SUMMARY:
The purpose of this study is to assess growth of preterm infants fed human milk supplemented with an experimental human milk fortifier.

ELIGIBILITY:
Inclusion Criteria:

* 700-1500g birth weight
* 33 weeks or less gestational age
* Appropriate for gestational age
* Initiate enteral feeds of human milk by 21 days of life
* Mother provided exclusive human milk feeds
* Parents allow both human milk and study human milk fortifier
* Singleton or twin birth

Exclusion Criteria:

* Feeding preterm infant formula or non-study human milk fortifier
* Expected at facility less than 15 days
* Congenital anomalies/disease affecting growth and development
* 5 minute APGAR of 4 or less
* Steroid use
* ECMO
* Grade III or IV PVH/IVH
* Mechanical ventilator dependency
* Maternal incapacity
* History of major surgery
* Asphyxia
* Confirmed NEC or sepsis
* Use of probiotics

Max Age: 21 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 147 (Actual)
Dates: Start 2011-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Weight gain | 29 days

SECONDARY OUTCOMES:
Anthropometric variables | 29 days
  Length and head circumference
GI tolerance | 29 days
  stool characteristics, periods of nil per os (NPO), and withheld feedings due to abdominal distention, gastric residuals, vomiting, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Bridget Barrett-Reis, PhD, Study Chair — Abbott Nutrition
Locations (15):
- United States (15):
  - University of Alabama, Birmingham, Alabama
  - UCSD Medical Center, San Diego, California
  - University South Florida, Tampa, Florida
  - Memorial Hospital of Southbend, Southbend, Indiana
  - Wesley Medical Center, Wichita, Kansas
  - King's County Hospital Center, Brooklyn, New York
  - Cohen Children's Medical Center of New York at North Shore, Manhasset, New York
  - Cohen Children's Medical Center of NY at North Shore, New Hyde Park, New York
  - Childrens Hospital Westchester Medical Center, Valhalla, New York
  - University Hospitals Case Medical Center Rainbow Babies & Children's Hospital, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Toledo Children's Hospital, Toledo, Ohio
  - OHSU, Portland, Oregon
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Kim JH, Chan G, Schanler R, Groh-Wargo S, Bloom B, Dimmit R, Williams L, Baggs G, Barrett-Reis B. Growth and Tolerance of Preterm Infants Fed a New Extensively Hydrolyzed Liquid Human Milk Fortifier. J Pediatr Gastroenterol Nutr. 2015 Dec;61(6):665-71. doi: 10.1097/MPG.0000000000001010. PMID 26488118